CLINICAL TRIAL: NCT02040779
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, 12-Week Clinical Study to Assess the Efficacy and Safety of Beclomethasone Dipropionate (80 and 160 mcg/Day) Delivered Via Breath-Actuated Inhaler (BAI) in Adolescent and Adult Patients 12 Years of Age and Older With Persistent Asthma
Brief Title: A 12-week Safety and Efficacy Study of Beclomethasone Dipropionate (80 and 160 mcg/Day) Delivered Via Breath-Actuated Inhaler (BAI) in Patients >=12 Years Old With Persistent Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BDB-AS-304
Record Dates: First submitted 2014-01-16; First posted 2014-01-20 (Estimated); Results first posted 2017-12-11 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Persistent Asthma
Keywords: asthma; breath-actuated inhaler; beclomethasone
MeSH Terms: conditions — Asthma | interventions — Albuterol; Bronchodilator Agents

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- BDP 80 mcg BAI (Experimental): 40 mcg beclomethasone dipropionate (BDP) via breath-actuated inhaler (BAI) twice daily for a total of 80 mcg/day.
  Interventions: Drug: Beclomethasone dipropionate breath-actuated inhaler; Drug: albuterol/salbutamol
- BDP 160 mcg BAI (Experimental): 80 mcg beclomethasone dipropionate (BDP) via breath-actuated inhaler (BAI) twice daily for a total of 160 mcg/day.
  Interventions: Drug: Beclomethasone dipropionate breath-actuated inhaler; Drug: albuterol/salbutamol
- Placebo BAI (Placebo Comparator): Placebo breath-actuated inhaler (BAI) twice daily.
  Interventions: Drug: Placebo breath-actuated inhaler; Drug: albuterol/salbutamol

INTERVENTIONS:
Drug: Beclomethasone dipropionate breath-actuated inhaler — Beclomethasone dipropionate (BDP) breath-actuated inhaler (BAI) given in dosages of either 40 mcg/inhalation or 80 mcg/inhalation. Study drug was administered twice each day, in the morning and in the evening, after the completion of the asthma symptom score and the PEF measurements, in that order.
  Other Names: BDP
  Arms: BDP 160 mcg BAI; BDP 80 mcg BAI
Drug: Placebo breath-actuated inhaler — Placebo was provided in matching breath-actuated inhaler (BAI) devices. The placebo devices were identical to the devices used to deliver active drug. Placebo was administered twice each day, in the morning and in the evening, after the completion of the asthma symptom score and the PEF measurements, in that order.
  Arms: Placebo BAI
Drug: albuterol/salbutamol — Rescue medication (albuterol/salbutamol hydrofluoroalkane (HFA) MDI [90 mcg ex-actuator] or equivalent) for use on an as-needed basis for the immediate relief of asthma symptoms throughout the treatment period
  Other Names: bronchodilators

SUMMARY:
This is a randomized, double-blind, placebo-controlled parallel-group study. Participants will be randomly assigned to receive treatment with beclomethasone dipropionate at a dosage of 80 or 160 mcg/day delivered via a Breath-Actuated Inhaler (BAI); or a matching BAI placebo, in a 1:1:1 ratio after a 14- to 21-day run-in period. Participants and investigators will remain blinded to randomized treatment assignment during the study

ELIGIBILITY:
Inclusion Criteria:

* Severity of Disease: The patient has persistent asthma, with an forced expiratory volume in 1 second (FEV1) 40%-85% of the value predicted for age, height, sex, and race as per the National Health and Nutrition Examination Survey (NHANES III) reference values at screening visit (SV) (Hankinson et al 1999).
* Current asthma therapy: The patient is currently being treated with 1 of the following:

  1) inhaled corticosteroids (ICSs) at a stable daily dose of less than or equal to 220 mcg/day fluticasone propionate via metered dose inhaler (MDI) or equivalent for a minimum of 4 weeks (28 days) before screening visit, or 2) a stable daily dosage of non-corticosteroid therapy, including leukotriene modifiers, theophylline, chromones, or short-acting beta-2 agonists (SABAs) alone or in combination for a minimum of 4 weeks (28 days) before screening visit (SV).
* Reversibility of disease: The patient has demonstrated at least 15% and at least 200 mL increase from baseline FEV1 (patients age 18 and older) within 30 minutes after 2-4 inhalations of albuterol/salbutamol hydrofluoroalkane (HFA) MDI (90 mcg ex-actuator) or equivalent at SV or on retesting. - Other criteria apply, please contact the investigator for more information

Exclusion Criteria:

* The patient has a history of life-threatening asthma, defined for this protocol as an asthma episode that required intubation and/or was associated with hypercapnea, respiratory arrest, or hypoxic seizures.
* The patient is a pregnant or lactating female or plans to become pregnant.
* The patient has a known hypersensitivity to any corticosteroid or any of the excipients in the study drug or rescue medication formulation.
* The patient currently smokes or has a smoking history of 10 pack-years or more (a pack-year is defined as smoking 1 pack of cigarettes/day for 1 year). The patient may not have used tobacco products within the past year.
* The patient has had an asthma exacerbation requiring oral corticosteroids within 1 month before SV, or has had any hospitalization for asthma within 2 months before SV.
* The patient has historical or current evidence of a clinically significant disease. Significant disease is defined as any disease that in the medical judgment of the investigator would put the safety of the patient at risk through participation or that could affect the efficacy or safety analysis if the disease/condition worsened during the study.
* Other criteria apply, please contact the investigator for more information

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2013-12-26; Primary Completion 2014-12-24 (Actual); Study Completion 2014-12-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (47):
- United States (47):
  - Teva Investigational Site 12813, Huntington Beach, California
  - Teva Investigational Site 10944, Mission Viejo, California
  - Teva Investigational Site 10946, Orange, California
  - Teva Investigational Site 10963, Rolling Hills Estates, California
  - Teva Investigational Site 10960, San Diego, California
  - Teva Investigational Site 10973, San Diego, California
  - Teva Investigational Site 10975, San Jose, California
  - Teva Investigational Site 10948, Centennial, Colorado
  - Teva Investigational Site 10958, Centennial, Colorado
  - Teva Investigational Site 10957, Colorado Springs, Colorado
  - Teva Investigational Site 12814, Sarasota, Florida
  - Teva Investigational Site 10962, Tallahassee, Florida
  - Teva Investigational Site 12809, Savannah, Georgia
  - Teva Investigational Site 10947, Indianapolis, Indiana
  - Teva Investigational Site 10943, Iowa City, Iowa
  - Teva Investigational Site 10954, Baltimore, Maryland
  - Teva Investigational Site 12940, Bethesda, Maryland
  - Teva Investigational Site 10955, North Dartmouth, Massachusetts
  - Teva Investigational Site 10941, Minneapolis, Minnesota
  - Teva Investigational Site 10970, Columbia, Missouri
  - Teva Investigational Site 10968, Rolla, Missouri
  - Teva Investigational Site 10972, Bozeman, Montana
  - Teva Investigational Site 12941, Missoula, Montana
  - Teva Investigational Site 10942, Bellevue, Nebraska
  - Teva Investigational Site 10959, Skillman, New Jersey
  - Teva Investigational Site 10945, Raleigh, North Carolina
  - Teva Investigational Site 12810, Cincinnati, Ohio
  - Teva Investigational Site 10974, Sylvania, Ohio
  - Teva Investigational Site 12805, Oklahoma City, Oklahoma
  - Teva Investigational Site 12942, Oklahoma City, Oklahoma
  - Teva Investigational Site 10951, Tulsa, Oklahoma
  - Teva Investigational Site 10940, Lake Oswego, Oregon
  - Teva Investigational Site 10952, Medford, Oregon
  - Teva Investigational Site 10956, Portland, Oregon
  - Teva Investigational Site 12939, Pittsburgh, Pennsylvania
  - Teva Investigational Site 12806, Orangeburg, South Carolina
  - Teva Investigational Site 12811, Knoxville, Tennessee
  - Teva Investigational Site 10969, Austin, Texas
  - Teva Investigational Site 12812, Boerne, Texas
  - Teva Investigational Site 10949, Dallas, Texas
  - Teva Investigational Site 10953, El Paso, Texas
  - Teva Investigational Site 12807, Houston, Texas
  - Teva Investigational Site 10950, New Braunfels, Texas
  - Teva Investigational Site 10961, San Antonio, Texas
  - Teva Investigational Site 12808, Waco, Texas
  - Teva Investigational Site 10967, Seattle, Washington
  - Teva Investigational Site 10964, Greenfield, Wisconsin

REFERENCES:
- [Derived] Hampel FC Jr, Carr W, Gillespie M, Small CJ. Evaluation of beclomethasone dipropionate (80 and 160 micrograms/day) delivered via a breath-actuated inhaler for persistent asthma. Allergy Asthma Proc. 2017 Nov 8;38(6):419-430. doi: 10.2500/aap.2017.38.4089. Epub 2017 Sep 8. PMID 28886758

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For this study, 47 sites were activated and screened at least 1 patient, 44 sites screened at least 1 patient who entered the run-in period, and 43 sites randomly assigned a patient. Overall, 273 patients were randomly assigned to treatment
Period: Overall Study
Arm/Group | Placebo BAI | BDP 80 mcg BAI | BDP 160 mcg BAI
Started | 91 | 90 | 92
Full Analysis Set (FAS) | 90 | 88 | 92
Completed | 79 | 83 | 88
Not Completed | 12 | 7 | 4
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 1 | 3
Not completed — Non-compliance | 0 | 1 | 0
Not completed — Protocol Violation | 2 | 1 | 0
Not completed — Lost to Follow-up | 1 | 2 | 1
Not completed — Lack of Efficacy | 4 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo BAI | BDP 80 mcg BAI | BDP 160 mcg BAI | Total
Number analyzed (Participants) | 91 | 90 | 92 | 273
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.2 (14.82) | 38.8 (15.02) | 37.4 (16.05) | 37.8 (15.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 54 | 56 | 156
  Male | 45 | 36 | 36 | 117
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 2 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 13 | 17 | 14 | 44
  White | 73 | 64 | 72 | 209
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 7 | 5 | 13
Weight [Mean (Standard Deviation); unit: kg] | 82.27 (23.848) | 85.30 (22.382) | 80.29 (20.577) | 82.60 (22.316)
Height [Mean (Standard Deviation); unit: cm] — Population: One participant did not have a height recorded
  cm
    number analyzed (Participants) | 90 | 90 | 92 | 272
    (all) | 169.28 (9.473) | 170.88 (10.447) | 168.78 (8.657) | 169.64 (9.554)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: One participant did not have a height recorded, therefore BMI could not be calculated.
  kg/m^2
    number analyzed (Participants) | 90 | 90 | 92 | 272
    (all) | 28.383 (6.9051) | 29.266 (7.9371) | 28.136 (6.7751) | 28.591 (7.2109)
Duration of Asthma [Count of Participants; unit: Participants]
  <3 months | 0 | 0 | 0 | 0
  3 months to <6 months | 0 | 1 | 0 | 1
  6 months to <1 year | 1 | 1 | 0 | 2
  1 year to < 5 years | 4 | 4 | 2 | 10
  5 years to <10 years | 9 | 8 | 10 | 27
  10 years to <15 years | 12 | 16 | 18 | 46
  >=15 years | 65 | 60 | 62 | 187
Current Asthma Therapy [Count of Participants; unit: Participants]
  Inhaled corticosteroid | 35 | 34 | 35 | 104
  Non-corticosteroid | 56 | 56 | 57 | 169

OUTCOME MEASURES:

1. Primary Outcome: Standardized Baseline-Adjusted Trough Morning Forced Expiratory Volume in One Minute (FEV1) Area Under the Effect Curve From Time Zero to 12 Weeks (AUEC(0-12wk)) by Actual Treatment Received
Description: The primary efficacy variable was the standardized baseline-adjusted trough morning (pre-dose and pre-rescue bronchodilator) FEV1 AUEC(0-12wk). Pulmonary function measurements such as FEV1 were obtained electronically by spirometry at the randomization visit (Day 1), each treatment visit (Weeks 2, 4, 8 and 12) and any unscheduled visit (such as the early termination visit). This summary is based on observed values recorded as 'best attempt'.
  The least-square (LS) means, difference of LS means and its 95% confidence interval (CI), and p-value represent the results obtained from the analysis of covariance with covariate adjustment for baseline, sex, age, current asthma therapy, and treatment.
Time Frame: Baseline (Day 1 predose), weeks 2, 4, 8 and 12
Population: The full analysis set (FAS) included all patients in the intent to treat (ITT) population who received at least 1 dose of study drug and had at least 1 postbaseline trough morning (pre-dose and pre-rescue bronchodilator) assessment of FEV1.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo BAI | BDP 80 mcg BAI | BDP 160 mcg BAI
Number analyzed (Participants) | 88 | 88 | 92
liters | 0.048 (0.0252) | 0.171 (0.0254) | 0.164 (0.0248)
Statistical Analysis 1: Comparison: Placebo BAI vs BDP 160 mcg BAI; A fixed-sequence multiple testing procedure was used while controlling the family-wise error rate at 5%. If the 2-sided p-value resulting from the ANCOVA model for comparing beclomethasone dipropionate BAI 160 mcg/day versus placebo was less than 0.05, then the comparison of the 80 mcg/day versus placebo was to be interpreted inferentially; Test type: Superiority; p = 0.0010, ANCOVA — ANCOVA model with effects due to baseline trough morning FEV1, sex, age, current protocol-allowed asthma therapy (ICS or non-corticosteroid therapy) at the time of screening visit and during the run-in period and treatment; LSM difference = 0.116, 95% CI 2-sided [0.048 to 0.185] — BDP 160 mcg BAI - Placebo BAI
Statistical Analysis 2: Comparison: Placebo BAI vs BDP 80 mcg BAI; Test type: Superiority; p = 0.0005, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LSM difference = 0.124, 95% CI 2-sided [0.054 to 0.193] — BDP 80 mcg BAI - Placebo BAI

2. Secondary Outcome: Change From Baseline in Weekly Average of Daily Trough Morning Peak Expiratory Flow (PEF) Rate Over the 12-Week Treatment Period
Description: Change from baseline in the weekly average of daily trough morning (pre-dose and pre-rescue bronchodilator) PEF by handheld spirometer over the 12-week treatment period.
  PEF were determined twice daily, in the morning and in the evening, before administration of study drug or rescue medications. A handheld spirometer was provided to patients and used to determine the morning and evening PEF throughout the study. The spirometer was programmed to record the highest PEF obtained from 3 valid attempts.
  Baseline was defined as the average of recorded trough morning PEF assessments over the 7 days prior to the first dose of double-blind study treatment, including the morning assessment at the randomization visit.
  The LS means, difference of LS means and its 95% confidence interval, and p value are obtained from the mixed model for repeated measures analysis with covariate adjustment for baseline, sex, age, current asthma therapy, treatment, week, and treatment by week interaction.
Time Frame: Baseline (Days -6 to Day 1 pre-dose), daily up to Week 12
Population: Full analysis set (FAS)
Measure: Least Squares Mean (Standard Error); unit: L/minute
Arm/Group | Placebo BAI | BDP 80 mcg BAI | BDP 160 mcg BAI
Number analyzed (Participants) | 89 | 88 | 92
L/minute | -0.795 (2.8224) | 12.849 (2.8241) | 7.116 (2.7735)
Statistical Analysis 1: Comparison: Placebo BAI vs BDP 160 mcg BAI; Treatment comparisons began with am PEF for BDP 160 mcg BAI vs placebo. If the p-value was ≤0.05, the next comparisons of interest were made 1) the next secondary outcome comparison for BDP 160 mcg BAI vs placebo and 2) the am PEF for BDP 80 mcg BAI vs placebo. This procedure allowed for control of the Type I error for comparisons at a particular BAI treatment over the 5 secondary endpoints, as well as comparisons within an endpoint. It did not control the overall Type I error; Test type: Superiority; p = 0.0443, mixed model for repeated measures — a priori threshold for significance of 0.05; LSM difference = 7.911, 95% CI 2-sided [0.202 to 15.621] — BDP 160 mcg BAI - Placebo BAI
Statistical Analysis 2: Comparison: Placebo BAI vs BDP 80 mcg BAI; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0007, mixed model for repeated measures — a priori threshold for significance of 0.05; LSM difference = 13.645, 95% CI 2-sided [5.843 to 21.446] — BDP 160 mcg BAI - Placebo BAI

3. Secondary Outcome: Change From Baseline in Weekly Average of Daily Evening Peak Expiratory Flow (PEF) Over the 12-Week Treatment Period
Description: A hand-held peak flow meter was provided to patients at the screening visit and used to determine the morning and evening PEF throughout the course of the study. The patient recorded the highest value of 3 measurements obtained in the morning and evening in the patient diary.
  Baseline in evening PEF is defined as the average of recorded evening PEF assessments over the 7-day window before randomization.
  The LS means, difference of LS means and its 95% confidence interval, and p value are obtained from the mixed model for repeated measures analysis with covariate adjustment for baseline, sex, age, current asthma therapy, treatment, week, and treatment by week interaction.
Time Frame: Baseline (Days -6 to Day 1 pre-dose), daily up to Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: L/minute
Arm/Group | Placebo BAI | BDP 80 mcg BAI | BDP 160 mcg BAI
Number analyzed (Participants) | 89 | 88 | 92
L/minute | -0.797 (3.0380) | 10.105 (35.0507) | 4.608 (2.9908)
Statistical Analysis 1: Comparison: Placebo BAI vs BDP 160 mcg BAI; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.2014, mixed model for repeated measures — a priori threshold for significance of 0.05; LSM difference = 5.405, 95% CI 2-sided [-2.905 to 13.715] — BDP 160 mcg BAI - Placebo BAI
Statistical Analysis 2: Comparison: Placebo BAI vs BDP 80 mcg BAI; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0112, mixed model for repeated measures — a priori threshold for significance of 0.05; LSM difference = 10.902, 95% CI 2-sided [2.500 to 19.303] — BDP 160 mcg BAI - Placebo BAI

4. Secondary Outcome: Change From Baseline in Weekly Average of Total Daily Use of Albuterol/Salbutamol Inhalation Aerosol Over Weeks 1-12
Description: Change from baseline in the use of rescue medication, albuterol/salbutamol, during the treatment period offers an indication of asthma control.
  The LS means, difference of LS means and its 95% CI, and p-value are obtained from the mixed model for repeated measures analysis with covariate adjustment for baseline, sex, age, current asthma therapy, treatment, week and treatment by week interaction.
  Baseline was defined as the average of recorded daily usage of albuterol/salbutamol inhalation aerosol over the 7 days prior to the first dose of double-blind study treatment, including morning usage at the randomization visit.
Time Frame: Baseline (Days -6 to Day 1 pre-dose), daily up to Week 12
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: inhalations
Arm/Group | Placebo BAI | BDP 80 mcg BAI | BDP 160 mcg BAI
Number analyzed (Participants) | 86 | 88 | 89
inhalations | -0.010 (0.1162) | -0.368 (0.1155) | -0.398 (0.1153)
Statistical Analysis 1: Comparison: Placebo BAI vs BDP 160 mcg BAI; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0175, mixed model for repeated measures — a priori threshold for significance of 0.05; LSM difference = -0.388, 95% CI 2-sided [-0.708 to -0.068] — BDP 160 mcg BAI - Placebo BAI
Statistical Analysis 2: Comparison: Placebo BAI vs BDP 80 mcg BAI; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0285, mixed model for repeated measures — a priori threshold for significance of 0.05; LSM difference = -0.358, 95% CI 2-sided [-0.678 to -0.038] — BDP 80 mcg BAI - Placebo BAI

5. Secondary Outcome: Change From Baseline in Weekly Average of Total Daily Asthma Symptom Score Over the 12-Week Treatment Period
Description: Asthma symptom scores were recorded in the patient's diary each morning and evening before determining FEV1 and PEF and before administration of study or rescue medications.
  The Daytime Symptom Score was recorded in the evening on a scale of 0 (No symptoms during the day) to 5 (Symptoms so severe that I could not go to work or perform normal daily activities) plus the Nighttime Symptom Score in the morning on a scale of 0 (No symptoms during the night) to 4 (Symptoms so severe that I did not sleep at all) for a total score range of 0-9.
  Baseline was defined as the average of recorded daily asthma symptom scores (average of daytime and nighttime score) over the 7 days prior to the first dose of study treatment, including the morning assessment at the randomization visit.
  The LS means, difference of LS means and its 95% CI, and p value are obtained from the mixed model for repeated measures analysis with covariate adjustment for baseline, sex, age, current asthma therapy,
Time Frame: Baseline (Days -6 to Day 1 pre-dose), daily up to Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo BAI | BDP 80 mcg BAI | BDP 160 mcg BAI
Number analyzed (Participants) | 90 | 88 | 92
units on a scale | -0.166 (0.0460) | -0.293 (0.0463) | -0.304 (0.0454)
Statistical Analysis 1: Comparison: Placebo BAI vs BDP 160 mcg BAI; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0335, mixed model for repeated measures — a priori threshold for significance of 0.05; LSM difference = -0.137, 95% CI 2-sided [-0.263 to -0.011] — BDP 160 mcg BAI - Placebo BAI
Statistical Analysis 2: Comparison: Placebo BAI vs BDP 80 mcg BAI; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0509, mixed model for repeated measures — a priori threshold for significance of 0.05; LSM difference = -0.127, 95% CI 2-sided [-0.255 to 0.001] — BDP 80 mcg BAI - Placebo BAI

6. Secondary Outcome: Kaplan-Meier Estimates of Time to Study Drug Treatment Withdrawal Due to Meeting Stopping Criteria for Worsening Asthma During the 12-Week Treatment Period
Description: The time to patient study drug treatment withdrawal due to worsening asthma was defined as the number of days elapsed from the date of randomization to the date of withdrawal due to meeting stopping criteria. Alert criteria for individual patients with worsening asthma were designed to ensure patient safety. The investigator determined whether the patient's overall clinical picture is consistent with worsening asthma and if the patient should be withdrawn from study drug treatment (but not the study) and be placed on appropriate asthma therapy in the interest of patient safety.
  An example of alert criteria is:
  * FEV1 as measured at the study center is below the FEV1 stability limit value calculated at randomization visit (Day 1).
  * Other criteria as defined in the protocol.
Time Frame: Treatment period: daily from Day 1 up to Week 12
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo BAI | BDP 80 mcg BAI | BDP 160 mcg BAI
Number analyzed (Participants) | 90 | 88 | 92
days | NA [NA to NA] — Insufficient number of participants withdrawn | NA [NA to NA] — Insufficient number of participants withdrawn | NA [NA to NA] — Insufficient number of participants withdrawn

7. Secondary Outcome: Number of Participants Withdrawn From Study Due to Meeting Stopping Criteria for Worsening Asthma During the 12-Week Treatment Period
Description: A count of participants who were withdrawn from the study due to meeting stopping criteria. Alert criteria for individual patients with worsening asthma were designed to ensure patient safety. The investigator determined whether the patient's overall clinical picture is consistent with worsening asthma and if the patient should be withdrawn from study drug treatment (but not the study) and be placed on appropriate asthma therapy in the interest of patient safety.
  An example of alert criteria is:
  * FEV1 as measured at the study center is below the FEV1 stability limit value calculated at randomization visit (Day 1).
  * Other criteria as defined in the protocol.
Time Frame: Treatment period: Day 1 up to Week 12
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo BAI | BDP 80 mcg BAI | BDP 160 mcg BAI
Number analyzed (Participants) | 90 | 88 | 92
Participants | 5 | 2 | 0
Statistical Analysis 1: Comparison: Placebo BAI vs BDP 80 mcg BAI; Test type: Superiority; p = 0.2384, Log Rank
Statistical Analysis 2: Comparison: Placebo BAI vs BDP 160 mcg BAI; Test type: Superiority; p = 0.0208, Log Rank

8. Secondary Outcome: Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Severity was rated by the investigator on a scale of mild, moderate and severe, with severe= an inability to carry out usual activities. Relation of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent 1 of the outcomes listed in this definition.
Time Frame: Day 1 up to Week 12
Population: The safety population included all randomly assigned patients (ITT population) who took 1 or more doses of study drug. In this population, treatment was assigned based upon the treatment patients actually received, regardless of the treatment to which they were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo BAI | BDP 80 mcg BAI | BDP 160 mcg BAI
Number analyzed (Participants) | 91 | 90 | 92
Participants
  >=1 adverse event | 28 | 32 | 26
  >=1 severe TEAE | 2 | 0 | 0
  >=1 treatment-related TEAE | 1 | 1 | 2
  >=1 serious TEAE | 1 | 0 | 0
  >=1 AE causing discontinuation | 1 | 0 | 0

9. Secondary Outcome: Participants With Potentially Clinically Relevant Abnormal Vital Sign Results During the Treatment Period
Description: Criteria for the select vital signs that showed a potentially clinically relevant abnormal result are:
  * Sitting systolic BP (low); <=90 mm Hg and decrease of >=20 mm Hg from baseline
  * Sitting diastolic BP (high): >=105 mm Hg and increase of >=15 mm Hg from baseline
  Baseline is defined as the last available assessment prior to the first dose of double-blind study treatment (usually Day 1 predose).
Time Frame: Baseline (Day 1 predose), Visits at weeks 2, 4, 8, 12
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo BAI | BDP 80 mcg BAI | BDP 160 mcg BAI
Number analyzed (Participants) | 91 | 90 | 92
Participants
  >=1 abnormality | 2 | 2 | 2
  Sitting systolic BP (low) | 1 | 1 | 1
  Sitting diastolic BP (high) | 1 | 1 | 1

10. Secondary Outcome: Participants With Findings During Oropharyngeal Examination During Treatment
Description: Oropharyngeal examinations were performed at every visit by a qualified healthcare professional: during treatment visits are summarized. Any visual evidence of oral candidiasis during the treatment period of the study was evaluated by obtaining and analyzing a swab of the suspect area for culturing. Appropriate therapy was to be initiated immediately at the discretion of the investigator and was not to be delayed for culture confirmation.
Time Frame: Visits at weeks 2, 4, 8, 12
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo BAI | BDP 80 mcg BAI | BDP 160 mcg BAI
Number analyzed (Participants) | 91 | 90 | 92
Participants
  >=1 evidence of oral candidiasis appearance | 0 | 0 | 2
  Participants with a positive culture | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Day 1 to Week 12
Arm/Group | Placebo BAI | BDP 80 mcg BAI | BDP 160 mcg BAI
All-Cause Mortality (participants affected / at risk) | 0/91 | 0/90 | 0/92
Serious Adverse Events (participants affected / at risk) | 1/91 | 0/90 | 0/92
Other Adverse Events (participants affected / at risk) | 0/91 | 0/90 | 0/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo BAI (N=91) | BDP 80 mcg BAI (N=90) | BDP 160 mcg BAI (N=92)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.